CLINICAL TRIAL: NCT01498315
Title: The Incidence of Pelvic Hematoma Following Hysterectomy
Acronym: Hematoma
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ron Auslender, Head of Obstetric and Gynecology, Carmel Medical Center
Other Study IDs: CMC-11-0073-CTIL
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Hematoma
MeSH Terms: conditions — Hematoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women following hysterecomy
  Interventions: Other: Ultrasound examination

INTERVENTIONS:
Other: Ultrasound examination — Ultrasound examination following hysterectomy

SUMMARY:
Hysterectomy is one of the common operations in gynecology. With population aging in modern society, the incidence of these surgeries is expected to increase even more. One of the major complications of pelvic surgery is symptomatic pelvic hematoma, which can present with pain, fever, and foul smelling discharge. The incidence of pelvic hematoma is 40%, and varies according to the type of hysterectomy and the diagnostic procedure. Those hematoma increase the risk for infection. Diagnosis usually is not a clinical one unless symptoms occur, and then the diagnosis is made by CT or ultrasound. Number of interventions are mentioned in the literature to try and decrease post operative complications and infections, none have suggested effective enough. This is a prospective study which objective is to characterize the incidence of pelvic hematoma following hysterectomy using ultrasound. The investigators will also try to identify preoperative, intraoperative and postoperative risk factors for infection of this hematomas. This identification might decrease the incidence of postoperative hematoma and infection.

DETAILED DESCRIPTION:
aging in modern society, the incidence of these surgeries is expected to increase even more. One of the major complications of pelvic surgery is symptomatic pelvic hematoma, which can present with pain, fever, and foul smelling discharge. The incidence of pelvic hematoma is 40%, and varies according to the type of hysterectomy and the diagnostic procedure. Those hematoma increase the risk for infection. Diagnosis usually is not a clinical one unless symptoms occur, and then the diagnosis is made by CT or ultrasound. Number of interventions are mentioned in the literature to try and decrease post operative complications and infections, none have suggested effective enough. This is a prospective study which objective is to characterize the incidence of pelvic hematoma following hysterectomy using ultrasound. The investigators will also try to identify preoperative, intraoperative and postoperative risk factors for infection of this hematomas. This identification might decrease the incidence of postoperative hematoma and infection.

ELIGIBILITY:
Inclusion Criteria:Women following Hysterectomy in the gynecologic division Carmel Medical Center

Exclusion Criteria:

* not relevant

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women following hysterectomy
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-03; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Inspection by Ultraspund of hematona | after hysterectomy
  Inspection by Ultraspund of hematona

CONTACTS AND LOCATIONS:
Overall Officials: Ron Auslender, Dr, Principal Investigator — Carmel Medical Center